CLINICAL TRIAL: NCT05742672
Title: Investigation of the Effect of Abdominal Massage Applied to Palliative Care Patients on Constipation and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Sevil PAMUK CEBECİ, Asst.Prof.Dr., Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-3
Record Dates: First submitted 2022-12-19; First posted 2023-02-24 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: MASSAGE
Keywords: Abdominal massage; Palliative care; Constipation; Quality of Life
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Massage (Experimental): In the experimental group, twice a day, in the morning and evening, and 30 minutes after the meal, for 15 minutes. Effusion, petrissage and vibration massage movements will be applied by the researcher for a certain period of time in accordance with the procedure (Abdominal Massage Application Directive). The application will continue for 7 days.
  Interventions: Other: ABDOMINAL MASSAGE APPLICATION

INTERVENTIONS:
Other: ABDOMINAL MASSAGE APPLICATION — * Experiment group twice a day in the morning and evening and 30 minutes after the feeding meal, for 15 minutes. For a period of time, effusion, petrissage, vibration massage movements will be applied by the researcher in accordance with the procedure (Abdominal Massage Application Directive). The application will continue for 7 days.- On the 3rd day (short term), 5th day (mid term) and 7th day (long term) to the massaged experimental group, the Constipation Severity Scale (CQS) and the Constipation Quality of Life Scale (QQQL) will be administered to determine the effect.
  * Day 7 Rome Ш Constipation Diagnostic Criteria (Annex: 2) will be applied again and the patient's constipation status will be evaluated for the last time.
  * Routine treatment and care practices in the clinic will continue.

SUMMARY:
The problem of constipation plays a very important role among these symptoms that patients experience intensely and negatively affect their quality of life. Although constipation is not a disease, it is a condition that causes discomfort to the person and may develop due to idiopathic reasons, as well as depending on diet, exercise habits, medications used and various disease processes. It may also occur. Constipation is one of the most common symptoms in patients treated in palliative care, and its prevalence is thought to be approximately 30-90%. Constipation is the third most common problem in palliative care, after pain and loss of appetite. Although drug therapy is the first method that comes to mind in the treatment of constipation, as it is known, medical treatment has many side effects risks and long-term drug use causes health problems. It creates a high financial burden on the care system. The high side effects and costs of laxative drugs used in the management of constipation necessitate the use of non-pharmacological methods. Non-pharmacological methods used in the management of constipation generally include regular exercise, fluid intake, and increased consumption of fiber foods. One of them is the abdominal massage method. The number of studies on the effects of abdominal massage in the Palliative Care patient group, who frequently experience constipation, is very limited in the literature. For these reasons, the study was planned to examine the effect of abdominal massage applied to palliative care patients on constipation and quality of life.

DETAILED DESCRIPTION:
The problem of constipation plays a very important role among these symptoms that patients experience intensely and negatively affect their quality of life. Although constipation is not a disease, it is a condition that causes discomfort to the person and may develop due to idiopathic reasons, as well as depending on diet, exercise habits, medications used and various disease processes. It may also occur. Constipation is one of the most common symptoms in patients treated in palliative care, and its prevalence is thought to be approximately 30-90%. Constipation is the third most common problem in palliative care, after pain and loss of appetite. Although drug therapy is the first method that comes to mind in the treatment of constipation, as it is known, medical treatment has many side effects risks and long-term drug use causes health problems. It creates a high financial burden on the care system. The high side effects and costs of laxative drugs used in the management of constipation necessitate the use of non-pharmacological methods. Non-pharmacological methods used in the management of constipation generally include regular exercise, fluid intake, and increased consumption of fiber foods. One of them is the abdominal massage method. The number of studies on the effects of abdominal massage in the Palliative Care patient group, who frequently experience constipation, is very limited in the literature. For these reasons, the study was planned to examine the effect of abdominal massage applied to palliative care patients on constipation and quality of life.Abdominal massage applied to palliative care patients It was planned in two stages to determine its effect on constipation and quality of life. The first phase of the study was descriptive and cross-sectional, and the second phase was planned as a randomized experimental study with a pretest-post test control group design.

In the first phase of the research, answers to the following questions will be sought.

What is the severity of constipation in palliative care patients?

-Performing daily living activities of palliative care patients How is the dependency independence situation?

Hypotheses of the Research:

H1: The application of abdominal massage to palliative care patients has an effect on constipation.

H1: The application of abdominal massage to palliative care patients has a positive effect on the quality of life.

The independent variable of the study was abdominal massage application, and the dependent variables were constipation and quality of life levels of palliative care patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the first phase of the study;
* A first-degree relative or volunteer to participate in the research approved to participate in the research by
* 18 years and over,
* Patients receiving inpatient treatment and care in the palliative care service. Inclusion criteria for the second phase of the study;
* A first-degree relative or volunteer to participate in the research approved to participate in the research by
* Having at least 2 or more of the Rome III constipation diagnostic criteria,
* Constipation Severity Scale score is 25 and above,
* No intestinal obstruction
* No radiotherapy or surgery was applied to the abdominal region until six weeks ago,
* Does not have diarrhea,
* Patients who do not have abdominal massage application restrictions.

Exclusion Criteria:

* Exclusion criteria for the first phase of the study;
* Those who do not volunteer to participate in the research or who are not approved to participate in the research by their first-degree relatives,
* under the age of 18,
* Patients who do not receive inpatient treatment and care in the palliative care service.

Exclusion criteria for the second phase of the study;

* Those who do not volunteer to participate in the research or who are not approved to participate in the research by their first-degree relatives,
* Below 2 of the Rome III constipation diagnostic criteria
* Constipation Severity Scale score below 25 points
* Intestinal obstruction
* Radiotherapy or surgery was applied to the abdominal region up to six weeks ago,
* Having diarrhea
* Patients with abdominal massage application restrictions will be formed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
To accept the hypothesis that the application of abdominal massage to palliative care patients has an effect on constipation. | 1 weeks
  Constipation Severity Scale (CSS) will be used to measure the effect of abdominal massage applied to the experimental group on constipation. There are 16 questions in the scale. The Constipation Severity Scale has three sub-dimensions: Stool Obstruction, Large Intestine Laziness, and Pain. The score that can be taken from the stool obstruction sub-dimension is 0-28, the score that can be taken from the large intestine laziness sub-dimension is between 0-29, and the score that can be taken from the pain sub-dimension is between 0-16. The lowest total score that can be obtained from the scale is 0, and the highest is 73. A high score on the scale indicates that the symptoms are serious.
To accept the hypothesis that the application of abdominal massage to palliative care patients has an impact on quality of life. | 1 weeks
  Constipation Quality of Life Scale, the scale developed to determine the effect of constipation on quality of life, consists of "worry/anxiety" (11 items), "physical discomfort" (4 items), "psychosocial discomfort" (8 items), "satisfaction" (5 items) subscales. consists of scales. The scale consists of 28 items in total. The highest score that can be obtained from the five-point Likert scale is 140, and the lowest score is 28. As the scores obtained from the scale increase, it is thought that the quality of life is negatively affected.

CONTACTS AND LOCATIONS:
Overall Officials: Sevil PAMUK CEBECİ, Asst.Prof., Study Director — sevil.pamukcebeci@ogu.edu.tr
Locations (2):
- Turkey (Türkiye) (2):
  - Sevil PAMUK CEBECİ, Eskişehir, Eskişehir
  - Eskişehir Şehir Hastanesi, Eskişehir

IPD SHARING:
Plan to Share IPD: No